CLINICAL TRIAL: NCT03485053
Title: 2 Part, Phase II Study of Intravenous, Single Ascending Dose Administrations of IOP Injection in Patients With Iron Deficient Anemia
Brief Title: A Single Ascending Study of IOP Injection in Patients With Iron Deficient Anemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor terminate the trial and will conduct a phase 2b clinical trial further
Sponsor: MegaPro Biomedical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IOP-CT-004
Record Dates: First submitted 2018-03-20; First posted 2018-04-02 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IOP Injection / MPB-1514 (Experimental): Administered IV infusion
  Interventions: Drug: IOP Injection / MPB-1514

INTERVENTIONS:
Drug: IOP Injection / MPB-1514 — Dilute with 5% Dextrose solution (D5W)

SUMMARY:
The purpose is to evaluate the efficacy and safety of IOP Injection (MPB-1514) for the treatment of iron-deficient anemia (IDA).

DETAILED DESCRIPTION:
The Phase II study is to establish the maximum tolerated dose of i.v. IOP Injection (MPB-1514) in Part 1 and to evaluate the safety and efficacy of the maximally tolerated dose of IOP Injection with different infusions schemes in Part 2.

ELIGIBILITY:
Inclusion Criteria:

1. Subject ≥ 18 years.
2. Subject with IDA but not secondary to any malignancy or renal failure requiring dialysis.
3. Hb levels <11.0 g/dL, Ferritin levels <200 ng/dL, Transferrin saturation (TSAT) < 20% at the Screening Visit.
4. Subject must have the ability to provide written, personally signed, and dated informed consent to participate in the study.
5. Subject must have an understanding, ability, and willingness to comply fully with study procedures and restrictions and to be available for clinic visits and follow-up procedures.
6. Female subject of child-bearing potential who is sexually active must use an effective method of birth control for at least one month prior to screening and agree to use an effective method of birth control until completion of participation in the study.

Exclusion Criteria:

1. Subject with known hemochromatosis, thalassemia, hemolytic anemia, receive red blood cell or whole blood transfusions within 90 days prior to enrollment.
2. Subject with a history of intravascular hemolysis.
3. Subject receiving any erythropoiesis-stimulating agent (ESA) therapy within 4 weeks prior to screenin.
4. Subject with a known sensitivity to any i.v. iron formulation
5. Subject with C-reactive protein > 20 mg/dL.
6. Subject with HBV, HCV, HIV.
7. Subject with known malignancy or severe renal failure requiring dialysis.
8. Subject with a recent (within 1 year of study drug administration) drug or alcohol abuse (including cannabis products) as defined in Diagnostic and Statistical Manual of Mental Disorders, 4th edition, Diagnostic Criteria for Drug and Alcohol Abuse.
9. Subject averages an intake of more than 21 units of alcohol per week (≥ 3 drinks per day) for men and 14 units of alcohol per week (≥ 2 drinks per day) for women (1 unit of alcohol equals approximately 250 mL of beer, 100 mL of wine or 35 mL of spirits).
10. Subject who has smoked or used smoking cessation or nicotine containing products (including but not limited to e-cigarettes, pipes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 6 months of the first dose of study drug.
11. Subject with any factor, which in the opinion of the Investigator would jeopardize the evaluation or safety or be associated with poor adherence to the protocol.
12. Subject with psychiatric disorder precluding the understanding of information on study related topics or giving informed consent.
13. Subject who has received another investigational agent within 4 weeks prior to screening.
14. Subject undergoing major surgery or physical trauma within 90 days or with major burn injury covering > 20% of total body surface area.
15. Female subject who is pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
The mean difference in Hb from baseline | on Day 28
  Evaluate in IDA patients by assessing changes in hemoglobin (Hb) levels after dosing

SECONDARY OUTCOMES:
The number of subjects with treatment-related serious adverse events | Day 0 to Day 28
  Safety will be assessed using the incidence of treatment-related serious adverse events
Pharmacokinetic analysis of IOP Injection: Peak Plasma Concentration | pre-dose to post-dose 24 hours
  Measurement of peak plasma concentration after dosing (Cmax)
Pharmacokinetic analysis of IOP Injection: Area Under the Plasma Concentration versus time | pre-dose to post-dose 24 hours
  Measurement of area under the plasma concentration versus time curve (AUC)
Pharmacokinetic analysis of IOP Injection: Half-life in Plasma | pre-dose to post-dose 24 hours
  Measurement of half-life of study drug in plasma after dosing (T1/2)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Fishbane, MD, Principal Investigator — North Shore University Hospital
Locations (8):
- United States (8):
  - North America Research Institute, Azusa, California
  - Valley Renal Medical Group, Northridge, California
  - Whittier Internal Medicine and Nephrology Medical Group, Whittier, California
  - South Florida Research Institute, Lauderdale Lakes, Florida
  - North Shore University Hospital Lab, Manhasset, New York
  - Clinical Research Development Associates, Springfield Gardens, New York
  - Northeast Clinical Research Center, Bethlehem, Pennsylvania
  - Southwest Houston Research Ltd., San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No